CLINICAL TRIAL: NCT04317157
Title: Placebo Effects and Physical Performance: Central and Peripheral Mechanisms Investigated by Different Experimental Designs
Brief Title: Placebo Effects Investigated by Different Experimental Designs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Principal Investigator, Flavio de Oliveira Pires, Head of Physical Activity Sciences Program, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: USP-NorthumbriaUNI
Record Dates: First submitted 2020-03-09; First posted 2020-03-23 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Caffeine; Placebo; Baseline
Keywords: Randomized clinical trial; Expectancy; Placebo; Caffeine
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: There are five experimental conditions in a crossover design. Participants will receive placebos in four of these trials and caffeine in the other one.
Who Masked: Participant, Investigator
Masking Description: Participants and the investigator that will be in touch with participants, will be blinded regarding the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Caffeine Clinical Trial (Experimental): Participants will ingest 6 mg.kg-1 of caffeine ~45 minutes before the trial, in a double-blinded, randomized clinical trial fashion.
  Interventions: Other: Placebo
- Placebo Clinical Trial (Placebo Comparator): Participants will ingest placebo ~45 minutes before the trial, in a double-blinded, randomized clinical trial fashion.
  Interventions: Other: Placebo
- Placebo-deceived Caffeine (Experimental): Participants will be lead to believe that they are ingesting 6 mg.kg-1 of caffeine ~45 minutes before the trial.
  Interventions: Other: Placebo
- Placebo-deceived Placebo (Placebo Comparator): Participants will be informed they are ingesting placebo ~45 minutes before the trial.
  Interventions: Other: Placebo
- Control-Caffeine (Active Comparator): Participants will be informed they are ingesting 6 mg.kg-1 of caffeine ~45 minutes before the trial.
  Interventions: Dietary Supplement: Caffeine
- Control (No Intervention): Participants will perform a baseline trial with no intervention.

INTERVENTIONS:
Dietary Supplement: Caffeine — Specific dosage of caffeine for each participant (6 mg.kg-1).
  Arms: Control-Caffeine
Other: Placebo — Placebo pill.
  Arms: Caffeine Clinical Trial; Placebo Clinical Trial; Placebo-deceived Caffeine; Placebo-deceived Placebo

SUMMARY:
This study aims to investigate the neurophysiological mechanisms of placebo perceived as caffeine during a motor task. Central and peripheral measures (i.e. electroencephalography and electromyography) will be assessed.

DETAILED DESCRIPTION:
Classical randomized clinical trial (RCT) controlled by a placebo is considered as the gold-standard design when evaluating the efficacy of drugs and interventions, as a given treatment is scientifically sound only if it is superior to placebo. One of strongest threats to placebo is that a double-blinded RCT could not completely neutralize every human consciousness-distorted reality; behavioral aspects such as the belief on a given treatment may directly result in different placebo effects and produce different treatment placebo effect sizes. Any patient may create his/her own expectation on a situation having a chance of 50% placebo vs 50% treatment depending on the available information; beliefs may impact on working mechanism of pharmacological treatments, but also on placebos. One alternative emerged from debates by different scientific fields; the control for the participant's expectancy by using an active substance-perceived placebo. When compared to a traditional double-blinded placebo-controlled RCT design, the placebo-deceived design has the advantage of controlling expectation and anxiety biases in treatments having combined pharmacological and psychological effects, despite some obvious limitation.

Mechanisms underpinning the ergogenic effect of placebos are unclear, but the suggestion is that the expectancy in using an ergogenic treatment/substance leads to psychobiological changes comparable to the actual treatment. A question that arises over RCT designs is how much effect on physical performance can be attributed to the actual substance and how much to the expectancy of receiving the actual substance. This question is relevant, as clinical and exercise settings have used double-blinded placebo-controlled RCT designs to investigate the ergogenic aids effects and mechanisms. However, participants may experience different placebo effect sizes in a double-blinded RCT design. This study will investigate ergogenic placebo effects and mechanisms elicited by double-blinded placebo-controlled RCT and deceived-placebo designs.

This crossover study will investigate two different experimental designs. During the traditional double-blind RCT, participants will be informed that they will be randomly assigned to caffeine and placebo sessions, thereby having 50% placebo chances vs 50% caffeine chances. However, they will receive placebo capsules in both RCT sessions (non-informed substance/received placebo). In contrast, they will be precisely informed about their allocation (either caffeine or placebo trial) in the deceived-placebo design, however they will ingest placebo capsules in both sessions (informed caffeine/received placebo vs informed placebo/received placebo), thereby controlling caffeine pharmacological effects. A true caffeine trial (informed caffeine/received caffeine 6 mg·kg-1) will be performed as a positive control in the last session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Must be able to swallow pills
* Must be able to perform isometric knee extension

Exclusion Criteria:

* Subjects with motor impairments

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Torque change | 30 minutes before the intervention and up to 60 minutes after the intervention
  Knee extension torque (N∙m) will be recorded during a maximal voluntary contraction through a load cell (EMG System ®, São José dos Campos, Brazil) coupled to a custom-built knee extension chair. Participants will have their torso individually adjusted on a backrest, in a comfortable position, fixed with straps to avoid body movement.
Rate of force development change | 30 minutes before the intervention and up to 60 minutes after the intervention
  Rate of force development (N∙m/s) will be recorded during a maximal voluntary contraction through a load cell (EMG System ®, São José dos Campos, Brazil) coupled to a custom-built knee extension chair. Participants will have their torso individually adjusted on a backrest, in a comfortable position, fixed with straps to avoid body movement.
Muscle activity change | Throughout the exercises performed 30 minutes before the intervention and up to 60 minutes after the intervention
  Vastus lateralis and vastus medialis muscles electromyography (EMG; (mV) will be assessed throughout both the exercises (maximal voluntary contraction and submaximal isometric voluntary contraction) according to standard recommendation.
H-reflex change | 30 minutes before the intervention and up to 60 minutes after the intervention
  H-reflex (mV) will be recorded at 10 s intervals through wireless electrodes placed over the vastus lateralis and vastus medialis muscles at rest, being considered as the peak-to-peak amplitude.
M-wave change | 30 minutes before the intervention and up to 60 minutes after the intervention
  M- and (mV) will be recorded at 10 s intervals through wireless electrodes placed over the vastus lateralis and vastus medialis muscles at rest, being considered as the peak-to-peak amplitude.
V-wave change | 30 minutes before the intervention and up to 60 minutes after the intervention
  V-wave (mV) and V-wave/Mmax (a.u.) will be recorded at 10 s intervals through wireless electrodes placed over the vastus lateralis and vastus medialis muscles at rest, being considered as the peak-to-peak amplitude.
Motor related cortical potential change | Throghout the isometric contraction 30 minutes before the intervention and up to 60 minutes after the intervention
  Will be recorded at Fz, Cz, Pz, C1 and C2 positions (µV) by using an electroencephalogram (EEG); the EEG recorded during the EMG burst (from 2 s before up to 4 s after the EMG onset) will be used to calculate the EEG amplitude (μv) in 4 windows within the muscle contraction such as; readiness potential (-1,5 to 0 s), muscle contraction 1 (0 to 1 s), muscle contraction 2 (1 to 2 s) and recovery (3 to 4 s).

SECONDARY OUTCOMES:
Ratings o perceived exertion change | Throughout the isometric contraction 30 minutes before the intervention and up to 60 minutes after the intervention
  Ratings of perceived exertion (RPE) will be obtained through a category-ratio (CR-10) Borg scale (u.a.). Participants will be familiarized with the scale anchors having the maximal voluntary contraction test as maximal effort template. The scale range from 0 - 10 reflecting the exerted effort (i.e. 0 for nothing at all and 10 extremely strong effort).

CONTACTS AND LOCATIONS:
Overall Officials: Flavio O Pires, Phd, Principal Investigator — School of Arts, Sciences and Humanities - University of São Paulo
Locations (1):
- School of Arts, Sciences and Humanities - University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Beedie C, Benedetti F, Barbiani D, Camerone E, Cohen E, Coleman D, Davis A, Elsworth-Edelsten C, Flowers E, Foad A, Harvey S, Hettinga F, Hurst P, Lane A, Lindheimer J, Raglin J, Roelands B, Schiphof-Godart L, Szabo A. Consensus statement on placebo effects in sports and exercise: The need for conceptual clarity, methodological rigour, and the elucidation of neurobiological mechanisms. Eur J Sport Sci. 2018 Nov;18(10):1383-1389. doi: 10.1080/17461391.2018.1496144. Epub 2018 Aug 16. PMID 30114971
- [Result] Pires FO, Dos Anjos CAS, Covolan RJM, Fontes EB, Noakes TD, St Clair Gibson A, Magalhaes FH, Ugrinowitsch C. Caffeine and Placebo Improved Maximal Exercise Performance Despite Unchanged Motor Cortex Activation and Greater Prefrontal Cortex Deoxygenation. Front Physiol. 2018 Aug 17;9:1144. doi: 10.3389/fphys.2018.01144. eCollection 2018. PMID 30246799